CLINICAL TRIAL: NCT00237133
Title: PREDICT TRIAL- Neoadjuvant Treatment of Locally Advanced Breast Cancer With Letrozole in Postmenopausal Women Expressing Hormonal Receptors ( ER and PR)
Brief Title: Treatment of Locally Advanced Breast Cancer With Letrozole in Postmenopausal Women
Acronym: PREDICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345EBR01
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Locally Advanced Breast Cancer
Keywords: Breast cancer,; Letrozole,; Hormonal receptors
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — 1 tablet of Letrozole 2.5 mg orally adminnistered once a day

SUMMARY:
Open-label Phase IV trial of Letrozole 2,5mg po/day for 120 days prior to surgery for patients with locally advanced breast in postmenopausal women expressing hormonal receptors ( ER and PR)

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women
2. Primary locally invasive breast cancer
3. Histological confirmed by core needle biopsy, whose tumors are estrogen (ER) and / or progesterone (PgR) positive, defined by core biopsy immunohistochemistry with > 10% positive malignant epithelial cells.
4. Post menopausal status
5. Tumor measurable by clinical examination, mammography and ultrasound

Exclusion Criteria:

1. Prior treatment with letrozole or tamoxifen.
2. Patients with bilateral breast tumors
3. Patients who are eligible for breast conserving surgery
4. Evidence of inflammatory breast cancer or distant metastasis.
5. Other concurrent malignant disease
6. Concomitant anti-cancer treatments such as chemotherapy

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2003-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Letrozole | frequency and severity of the clinical adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Brazil (11):
  - Novartis Investigative Site, Barretos - SP
  - Novartis Investigative Site, Florianopolis - SC
  - Novartis Investigative Site, Fortaleza/CE
  - Novartis Investigative Site, Goiania/GO
  - Novartis Investigative Site, Jau -SP
  - Novartis Investigative Site, Porto Alegre/RS
  - Novartis Investigative Site, Ribeirao - SP
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Santo André
  - Novartis Investigative Site, Sao Paulo/SP
  - Novartis Investigative Site, Vitoria/ES